CLINICAL TRIAL: NCT05676567
Title: Golf After Orthopaedic Surgery: A Longitudinal Follow-up (GOLF) Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 305142
Record Dates: First submitted 2022-12-20; First posted 2023-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis; Shoulder Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hip Arthroplasty: Patients undergoing total hip replacement, hip resurfacing or revision hip replacement
- Knee Arthroplasty: Patients undergoing total knee replacement, partial knee replacement or revision knee replacement
- Shoulder Arthroplasty: Patients undergoing total shoulder replacement, reverse shoulder replacement or partial shoulder replacement (hemiarthroplasty).

SUMMARY:
Aims The primary aim of this prospective, multi-centre study is to describe the rates of returning to golf following hip, knee and shoulder arthroplasty in an active golfing population. Secondary aims will include determining the timing of return to golf, changes in ability, handicap, and mobility, and assessing joint-specific and health-related outcomes following surgery.

Methods This is a multi-centre, prospective, longitudinal study between the Hospital for Special Surgery, New York City and Edinburgh Orthopaedics, Royal Infirmary of Edinburgh, United Kingdom. Both centres are high-volume arthroplasty centres, specialising in upper and lower limb arthroplasty. Patients undergoing hip, knee or shoulder arthroplasty at either centres, and who report being golfers prior to arthroplasty will be included. Patient-reported outcome measures will obtained at 6 weeks, 3 months, 6 months and 12 months. A one-year period of recruitment will be undertaken of arthroplasty patients at both sites.

Conclusions The results of this prospective study will provide clinicians with accurate data to deliver to patients with regards to the likelihood of return to golf and timing of when they can expect to return to golf following their hip, knee or shoulder arthroplasty, as well as their joint-specific functional outcomes. This will help patients to manage their postoperative expectations and plan their postoperative recovery pathway.

DETAILED DESCRIPTION:
This study will include adult patients who participate in golf (>18 years) at the Trauma and Orthopaedic Surgery Department, The Royal Infirmary of Edinburgh;) undergoing joint arthroplasty. The study will commence once NHS research ethics committee (REC) approval and NHS R&D Management approval is granted at the Royal Infirmary of Edinburgh.

The treatment that patients receive will not be affected by involvement in the study. The only difference in the patient pathway will be additional phone call/online follow ups of golf-related outcome measures postoperatively.

All patients will be identified in the clinic or pre-assessment clinic by the surgical team (consultant or registrar) or research assistant and be given the patient information sheet at one of these visits. Patients undergoing joint replacement in the orthopaedic unit are already offered to consent to follow up in the arthroplasty database at the time of attending the pre-assessment clinic and therefore additional paperwork will be added to enrol in the proposed golf study.

Patients will have access to the consent form at either the clinic or pre-assessment clinic. They are routinely offered to consent for arthroplasty follow up via our database which is in the form of 6 and 12 month postal questionnaires. An additional consent form will be included if patients identify as golfers on the questionnaire at the time of consenting for routine their arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years 2. A self-reported golfer 3. Able to consent to treatment 4. Assessed and listed for one of the following surgical procedures

  1. Total hip arthroplasty
  2. Hip resurfacing
  3. Revision hip arthroplasty
  4. Total knee arthroplasty
  5. Unicompartmental knee arthroplasty
  6. Revision knee arthroplasty
  7. Total shoulder arthroplasty
  8. Reverse shoulder arthroplasty
  9. Shoulder resurfacing arthroplasty
  10. Revision shoulder arthroplasty

Exclusion Criteria:

* 1. Patients unable to comply with post-operative data gathering including completing questionnaires 2. Patients declining operative management 3. No desire to return to golf postoperatively 4. Medical co-morbidities that affect the patient's ability to play golf, that will ultimately not allow the patient to return to golf postoperatively

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients scheduled for hip, knee and shoulder arthroplasty at each centre will be asked if they consider themselves a golfer. Potential patients will include those undergoing hip, knee or shoulder arthroplasty at the two medical centres. Patients will be enrolled preoperatively and followed for 1 year postoperatively.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate and timing of returning to golf following hip, knee and shoulder arthroplasty | 1 year
  The primary outcome will be to report the rates of return to golf following hip, knee and shoulder arthroplasty.

SECONDARY OUTCOMES:
Golf related outcomes | 1 year
  Secondary outcomes will include the timing of return, changes in the frequency of golfing, changes in mobility on the golf course, changes in handicap, joint pain during and after golf, and satisfaction with their involvement in golf.
Patient-reported outcome measure 1 | 1 year
  Golf After Arthroplasty Surgery Score
Patient-reported outcome measure 2 | 1 year
  Hip Disability and Osteoarthritis Outcome Score - Joint Replacement (HOOS-JR)
Patient-reported outcome measure 3 | 1 year
  Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS-JR)
Patient-reported outcome measure 4 | 1 year
  American Shoulder and Elbow Score (ASES)
Patient-reported outcome measure 5 | 1 year
  PROMIS Global Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Edinburgh Orthopaedics, Edinburgh, Midlothian, United Kingdom